CLINICAL TRIAL: NCT07366151
Title: The Impact of Active Screening on the Long-term Health of Celiac Disease Patients and the Natural Course of Potential Untreated or Treated Celiac Disease
Brief Title: Long-term Health Outcomes of Screen Detected and Potential Celiac Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Finnish Medical Foundation (Network)
Responsible Party: Sponsor
Other Study IDs: R24071
Record Dates: First submitted 2025-05-02; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Disease; Digestive System Diseases; Celiac Disease
Keywords: Celiac disease; Potential celiac disease; Gluten-free diet; Screen detected; Long-term health; Quality of life; Symptoms; Asymptomatic
MeSH Terms: conditions — Malabsorption Syndromes; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Duodenal mucosal biopsies, mucosal samples (oral cavity), stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screen detected CeD: Patients with confirmed celiac disease diagnosis found by screening of the disease
- Potential CeD: Patients earlier diagnosed with potential celiac disease and patients who have had celiac disease antibody positivity, but were not investigated further. Current diagnostic and treatment status is mostly unknown.

SUMMARY:
The primary aim of this project is to investigate how active screening and the timing of diagnosis affect the long-term health outcomes of patients with celiac disease. Additionally, the study seeks to clarify the natural course of so-called potential celiac disease. A key focus is also placed on assessing adherence to a gluten-free diet among screen-detected and, if initiated, potential celiac disease patients, their satisfaction with the diagnosis, and the diet's impact on general health and quality of life.

DETAILED DESCRIPTION:
In this retrospective observational cohort study, participants from earlier studies conducted by the Tampere Celiac Disease Research Center are invited for a follow-up visit. The study cohorts include individuals with screen-detected celiac disease (CeD), potential CeD, and subjects previously investigated due to positive CeD serology, but with an unknown diagnostic status. The participants are interviewed and complete structured questionnaires. Blood, urine, stool, and mucosal samples are collected for both routine clinical assessment and research purposes. Bone mineral density is measured using DXA, and a skin biopsy is offered to assess for latent dermatitis herpetiformis. Esophagogastroduodenoscopy is offered to participants with potential CeD who are on a gluten-containing diet, as well as to those experiencing challenges with dietary treatment. Clinical results are compared with healthy relatives and previously studied, treated CeD controls.

ELIGIBILITY:
Inclusion Criteria:

* Finnish citizenship and current residence in Finland

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of earlier study cohorts investigating potential or screen-detected celiac disease, irrespective of the current diagnostical status.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptom rating scale (GSRS) | At the time of study visit
  Symptoms are measured with Gastrointestinal symptom rating scale (GSRS) questionnaire. The scoring consists of 15 items, which are scored with a 7-grade Likert scale in which 1 point indicates no symptoms and 7 points the most severe gastrointestinal symptoms. Items cover five different symptoms (indigestion, diarrhea, abdominal pain, constipation and reflux) and values for each sub-dimension are calculated as a mean of the relevant items. The total GSRS score is described as a mean value of all 15 items (from 1 to 7 points). Scores of the participants are compared with the result of earlier study when possible.
Quality of life (PGWB) | At the time of study visit
  Quality of life is measured with Psychological General Well-Being (PGWB) questionnaire. The survey consists of 22 separate items covering six different sub-dimensions: anxiety, depression, well-being, self-control, general health and vitality. The scoring is based on a 6-grade Likert scale in which higher scores indicate better quality of life. The value of the total PGWB score may range from a minimum of 22 to maximum 132. The sub-scores are calculated as a sum of the items in each sub-dimensio. The PGWB results are compared with the result of earlier study when possible.

SECONDARY OUTCOMES:
Celiac disease diagnosis | 2-20 years
  How many have received celiac disease diagnosis after previous study?
Gluten-free diet | The time of study visit
  Adherence to the dietary treatment, when initiated is assessed by food diaries and Celiac Disease Adherence Test (CDAT) questionnaire. CDAT questionnaire is a 7-item questionnaire. Scoring is from 7 to 35, in which lower scores indicate good adherence and higher scores point towards poor adherence to gluten-free diet.
Skin symptoms | At the time of study visit
  Interview and Dermatology Life Quality Index (DLQI) questionnaire. The DLQI is dermatology-spesific index with 10 questonnaire considering the impact of skin disease to quality of life during the last week. Each question is scored with a 4-point Likert scale (0-3), giving the total DLQI score from 0 to 30, a higher score indicating worse quality of life
BMI | At the time of the study
  Weight (kilograms) and height (centimeters) will be combined as body mass index, kg/m2
Nutritional status and general health | 2-20 years
  Interview and blood tests
Bone mineral density | At the time of the study visit
  Bone mineral density is assessed with Duel-energy WX-ray Absorptiometry (DXA). In DXA, T-score compares bone mineral density to values of young, healthy adult. T-score -2.5 or lower indicates osteoporosis and score between -1.0 and -2.4 indicates osteopenia.
Modified Marsh-Oberhuber Classification | 2-20 years
  Duodenal histology is evaluated with morphological description and Modified Marsh-Oberhuber classification. In this classification Marsh 0 means entirely normal mucosa, Marsh 1 indicates normal villi and crypts with increased intraepithelial lymphocytes (IEL), Marsh 2 for increased IELs and crypt hyperplasia. Marsh 3 a-c villus atrophy is combined to increased IELs and cryp hyperplasia: Class 3a partial villus atrophy, 3b for subtotal villus atrophy and 3c for total villus atrophy.
Villus hight-Crypt depth Ratio (Vh/CrD) | 2-20 years
  Vh/CrD is a morphometric method to assess duodenal histology in addition to classifications like Marsh-Oberhuber. From several well-oriented duodenal samples, villous hight and crypt depth are measured. Ratio <2.0 indicates active celiac disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University, Faculty of Medicine and Health Technology, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No